CLINICAL TRIAL: NCT02595710
Title: Undetected Bartonella Spp. Infection Puts Liver Transplant Patients at Great Risk
Brief Title: Bartonella in Liver Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1312m46162
Record Dates: First submitted 2015-10-19; First posted 2015-11-03 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Cryptogenic Cirrhosis; Cryptogenic Chronic Hepatitis
Keywords: Cryptogenic Chronic Hepatitis; Bartonellosis
MeSH Terms: conditions — Cirrhosis, Cryptogenic; Hepatitis, Chronic; Bartonella Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Alpha Proteobacterium Growth Medium (BAPGM) multi-platform testing, including liquid culture, enriched agar plating and molecular techniques. Four-mm skin biopsies from non-lesional skin will be acquired from the same patients, processed using our published techniques, and imaged using confocal microscopy and compared to BAPGM test results. Urine samples will be collected and analyzed for microRNAs. Blood smears will be analyzed for intra-erythrocytic Bartonella spp.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biospecimen retention: Blood Collection Skin Punch Biopsy Collection Urine Sample Collection
  Interventions: Other: skin punch biopsy collection; Other: Blood collection; Other: Urine sample collection

INTERVENTIONS:
Other: skin punch biopsy collection — Four-mm skin biopsies from non-lesional skin will be acquired from the patients, processed using our published techniques with Bartonella biomarkers, and imaged using confocal microscopy.
Other: Blood collection — Blood will be tested for presence of Bartonella DNA and Bartonella antibodies using the Alpha Proteobacterium Growth Medium (BAPGM) multi-platform testing, including liquid culture, enriched agar plating and molecular techniques.Blood smears will be analyzed for presence of intra-erythrocytic Bartonella spp. by immunostaining.
Other: Urine sample collection — Urine samples will be collected and analyzed for Bartonella spp specific microRNAs.

SUMMARY:
Approximately 20 volunteers who have received a liver transplant and have been diagnosed with cryptogenic cirrhosis will be included in this study. Blood, skin and urine samples will be analyzed for Bartonella spp..

DETAILED DESCRIPTION:
Approximately 20 volunteers who have received a liver transplant and have been diagnosed with cryptogenic cirrhosis will be included in this study. Blood samples will be analyzed for Bartonella using the state-of-the art Bartonella Alpha Proteobacterium Growth Medium (BAPGM) multi-platform testing, including liquid culture, enriched agar plating and molecular techniques. Blood smears will be analyzed for intra-erythrocytic Bartonella spp. Four-millimeter skin biopsies from non-lesional skin will be acquired from the same patients, processed using our published techniques, and imaged using confocal microscopy and compared to BAPGM test results. additionally, urine samples will be collected and analyzed for microRNAs.

ELIGIBILITY:
Inclusion Criteria:

* o Male and female subjects, ages 18 years and older

  * Liver transplant recipient
  * Diagnosis of cryptogenic cirrhosis
  * Signed consent form

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes subjects ages 18 and above. Patients of the University of Minnesota Transplant Center who meet the inclusion/exclusion criteria will be given the opportunity to participate in this study. Dr. Lake has several liver transplant clinics and appropriate patients will be offered the opportunity to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Liver transplant subject that show evidence of Bartonella DNA and Bartonella antibodies using the Alpha Proteobacterium Growth Medium (BAPGM) | 90 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marna E Ericson, phd, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share individual patient data (IPD) with other researchers upon requet.